CLINICAL TRIAL: NCT00305916
Title: Accuracy of Multislice Spiral Computed Tomography in Diagnosis of Coronary Artery Disease Associated to Idiopathic Cardiomyopathy in Sinus Rhythm ("MSCT-IC Study").
Brief Title: Multislice Spiral Computed Tomography and Cardiomyopathy
Acronym: CMD-scanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Direction of Clinical Research and Strategy, Rennes University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AFSSAPS 2005/06/004; CIC0203/045; LOC/04-05
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2008-02

CONDITIONS: Cardiomyopathies
Keywords: MSCT; Idiopathic Cardiomyopathy; Sinus rhythm
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): conventional coronary angiography
  Interventions: Procedure: conventional coronary angiography
- 2 (Experimental): multislice spiral computed tomography coronary angiography
  Interventions: Procedure: Multislice spiral computed tomography coronary angiography

INTERVENTIONS:
Procedure: Multislice spiral computed tomography coronary angiography
  Other Names: MSCT
  Arms: 2
Procedure: conventional coronary angiography
  Arms: 1

SUMMARY:
Conventional coronary angiography is the recommended procedure in detection of coronary stenosis in patients with idiopathic cardiomyopathy. The aim of this prospective study is to assess diagnostic accuracy of multislice spiral computed tomography coronary angiography in patients with idiopathic cardiomyopathy in sinus rhythm, compared to conventional coronary angiography.

DETAILED DESCRIPTION:
The principal aim of this study is to assess the diagnostic accuracy (sensitivity, specificity, predictive values) of multislice spiral computed tomography (MSCT) coronary angiography among patients having idiopathic hypokinetic dilated cardiomyopathy in sinus rhythm, compared to conventional coronary angiography. The secondary aims are to assess the performance of MSCT in coronary sinus anatomy assessment, and in quantitative measurement of left ventricular anatomical criteria (telediastolic diameter, septal and posterior wall thickness, and ejection fraction) compared to echocardiography. Lastly, renal tolerance of MSCT will be studied. This prospective monocentric study will include 120 patients scheduled to undergo coronary angiography for etiologic diagnosis of idiopathic cardiomyopathy (defined by a left ventricle echographic ejection fraction ≤ 40 %, without anamnestic or electrocardiographic arguments in favour of coronary artery disease) in sinus rhythm. MSCT will be performed within 3 months after conventional coronary angiography, with blinded analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo coronary angiography,
* etiologic diagnosis of idiopathic cardiomyopathy (defined by a left ventricle echographic ejection fraction ≤ 40 %, without anamnestic or electrocardiographic arguments in favour of coronary artery disease),
* in sinus rhythm,
* informed written consent.

Exclusion Criteria:

* allergy to iodine,
* history of coronary artery bypass graft,
* history of percutaneous coronary angioplasty,
* history of myocardial infarction,
* known coronary artery disease,
* Q waves on the ECG,
* unstable haemodynamic status,
* urgent revascularisation or urgent valvular surgery,
* heart rate > 80 bpm (before MSCT),
* pregnancy,
* enrollment in another study.
* severe renal or respiratory insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Detection of > 50% coronary stenosis | During assessment
Sensibility, specificity, positive and negative predictive values of MSCT | During assessment

SECONDARY OUTCOMES:
Detection of patients with one or more coronary stenosis | During assessment
Detection of patients with 3-vessel disease | During assessment
Left ventricle telediastolic diameter | During assessment
Septal telediastolic thickness | During assessment
Posterior wall telediastolic thickness | During assessment
Detection of coronary sinus branches | During assessment
Measurement of coronary sinus branches diameter | During assessment
Assessment of renal function 7 days after MSCT | During assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Boulmier, MD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital; David Veillard, MD, Study Chair — Rennes University Hospital
Locations (1):
- Unité Fonctionnelle d'Hémodynamique et Cardiologie Interventionnelle - Hôpital Pontchaillou, Rennes, France